CLINICAL TRIAL: NCT05313516
Title: OKKO Space Academy App: Families Checking Their Child's Vision at Home During Amblyopia Treatment
Brief Title: OKKO Space Academy to Check Children's Vision at Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DALA1052
Record Dates: First submitted 2021-12-01; First posted 2022-04-06 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OKKO Health app (Experimental): Use of OKKO Health app for home monitoring.
  Interventions: Device: OKKO Health app

INTERVENTIONS:
Device: OKKO Health app — Use of OKKO Health app for home monitoring.

SUMMARY:
The purpose of this study is to determine the feasibility of the OKKO Space Academy app as a vision measuring and home-monitoring tool for children aged 3-8 years undergoing amblyopia treatment.

There are three objectives to this work:

1. Determine the feasibility of the OKKO Space Academy app for use between clinic visits from the child's and family perspective (i.e., acceptability, usability and engagement).
2. Assess the variability in day-to-day OKKO Health measurements between clinic visits (e.g., do the interim OKKO home vision measurements predict improvements in visual acuity?)
3. Explore agreement between the OKKO Space Academy measures of visual acuity against in-clinic measurements (usual standard of care), including an exploration of intra- and inter-session repeatability.

ELIGIBILITY:
Inclusion Criteria:

* Age 3.01 - 8.99 years with amblyopia
* Currently undergoing or at first visit to start amblyopia patching treatment
* Vision is fully corrected in glasses
* Visual acuity between -0.02 and 0.98 logMAR
* Have daily access to an approved smartphone or tablet
* Parent/child able to read and understand English
* Patient (child) able to understand spoken English

Exclusion Criteria:

* Parent not able to read and understand English
* Patient (child) not able to understand spoken English
* Parent/child not willing to participate
* Parent unable to give consent
* Any other ocular comorbidities
* Child has cognitive impairment or intellectual disability

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-06-26 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of home monitoring using the OKKO Health app | 3 months
  The feasibility and acceptability of the OKKO Space Academy app for use between clinic visits from the child's and family perspective. This will be assessed through a purpose built questionnaire.
Engagement of home monitoring using the OKKO Health app | 3 months
  The rate of engagement with the OKKO Space Academy app for use between clinic visits by the child (patient) and the family.
Variability in app data. | 3 months
  The variability in day-to-day OKKO Health measurements between clinic visits (e.g., do the interim OKKO home vision measurements predict changes in visual acuity?)
Visual acuity | 3 months
  Exploring the agreement between the OKKO Space Academy measures of visual acuity against in-clinic measurements (usual standard of care), including an exploration of intra- and inter-session repeatability.

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom